CLINICAL TRIAL: NCT05981976
Title: A Randomized, Open-Label, Parallel-Group, Single-dose, Relative Bioavailability Study of the Pharmacokinetics of Subcutaneous Abatacept (BMS-188667) Drug Product Converted From Drug Substance of a New Abatacept Drug Substance Process J Relative to the Current Abatacept Drug Process F in Healthy Participants
Brief Title: A Study to Evaluate the Drug Levels of Abatacept Converted From Drug Substance by Two Different Processes in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-920
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
Keywords: Abatacept; Orencia; Pharmacokinetics; Bioavailability; BMS-188667
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abatacept Treatment A (Experimental)
  Interventions: Biological: Abatacept
- Abatacept Treatment B (Experimental)
  Interventions: Biological: Abatacept

INTERVENTIONS:
Biological: Abatacept — Specified dose on specified days
  Other Names: Orencia®; BMS-188667

SUMMARY:
The purpose of this study is to compare the relative absorption of abatacept in healthy participants following subcutaneous (SC) administration in which the drug substance is manufactured with the current or new process.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, defined as having no clinically significant deviation from normal in medical history; physical examinations that would compromise the ability to participate, complete, and/or interpret the results of the study; 12-lead ECG; vital signs; and clinical laboratory results
* Body weight between 60 and 100 kilograms (kg) inclusive, based on weight at screening
* Participant must have a suitable injection site without tattoos, scarring, or other conditions in the upper, outer arm that could interfere with SC administration

Exclusion Criteria:

* Present malignancy or previous malignancy within the last 5 years prior to screening
* At risk for tuberculosis
* Any chronic bacterial infection within the previous 12 weeks of dosing

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to Day 71
Area under the serum concentration-time curve from time zero to the last time of quantifiable concentration (AUC(0-T)) | Up to Day 71
Area under the serum concentration-time curve from time zero extrapolated to infinity (AUC(INF)) | Up to Day 71

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Month 12
Number of participants with clinical laboratory abnormalities | Up to Month 12
Number of participants with vital sign abnormalities | Up to Month 12
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 71
Area under the serum concentration-time curve from time zero to 168 hours after dosing (AUC(0-168 hours)) | Up to Day 71
Serum concentration at 168 hours after dosing (C168) | Up to Day 71
Time of maximum observed serum concentration (Tmax) | Up to Day 71
Number of laboratory-reported positive responses of anti-abatacept antibodies | Up to Month 12
Number of laboratory-reported positive responses of anti-CTLA4-T antibodies | Up to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution, Cypress, California
  - Local Institution, Miami, Florida
  - Local Institution, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT05981976.html